CLINICAL TRIAL: NCT02616302
Title: A Phase 2, Double-Blind, 12-Week, Multicenter Study to Assess the Safety and Effectiveness of Daily Oral Administration of Dexlansoprazole Delayed-Release Capsules in Pediatric Subjects Aged 2 to 11 Years With Symptomatic Nonerosive Gastroesophageal Reflux Disease
Brief Title: A Study to Check the Safety of Dexlansoprazole and Learn if it Can Treat Symptomatic Nonerosive Gastroesophageal Reflux Disease in Children 2 to 11 Years Old
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-390MR_204; 2022-501349-64-00 (EU CTIS Number: EU CTIS); U1111-1166-8748 (Registry Identifier: WHO)
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Drug therapy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Weight ≤30 kg: Dexlansoprazole 15 mg (Experimental): Dexlansoprazole 15 mg, capsules, once, daily, for 12 weeks. Participants weigh ≤30 kg.
  Interventions: Drug: Dexlansoprazole
- Weight ≤30 kg: Dexlansoprazole 30 mg (Experimental): Dexlansoprazole 30 mg, capsules, once, daily, for 12 weeks. Participants weigh ≤30 kg.
  Interventions: Drug: Dexlansoprazole
- Weight >30 kg: Dexlansoprazole 30 mg (Experimental): Dexlansoprazole 30 mg, capsules, once, daily, for 12 weeks. Participants weigh >30 kg.
  Interventions: Drug: Dexlansoprazole
- Weight >30 kg: Dexlansoprazole 60 mg (Experimental): Dexlansoprazole 60 mg, capsules, once, daily, for 12 weeks. Participants weigh >30 kg.
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole 15 mg, 30 mg, and 60 mg capsules
  Other Names: Dexilant

SUMMARY:
Gastroesophageal reflux disease (GERD) is caused by food or acid coming up from the stomach into the esophagus, repeatedly. The esophagus is the tube that carries food and liquids from the mouth to the stomach.

The body uses stomach acid to break down food, but when acid rises up into the esophagus it can hurt or damage it. People with GERD often feel food coming back up into the throat and mouth and have a burning feeling in their stomach, chest, or throat, called heartburn. Other symptoms of GERD include pain in the stomach or throat, difficulty eating, and throwing up. Symptomatic nonerosive GERD is a condition where people have the symptoms of GERD but the esophagus has not been damaged. People of all ages can have GERD. The causes of GERD in children are similar to those in adults and teenagers.

Dexlansoprazole is a medicine that has been shown to help relieve the symptoms of GERD in adults and teenagers. This study aims to find out if dexlansoprazole doses given to children with symptomatic nonerosive GERD, based on their body weight, helps them feel better.

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. Dexlansoprazole is being tested to treat children aged 2 to 11 years who have nonerosive GERD. This study will look at the effectiveness and side effects of three different doses of dexlansoprazole in children with GERD.

The study will enroll approximately 70 patients. Participants weighing ≤30 kilograms (kg) will be randomly assigned (by chance, like flipping a coin) to receive dexlansoprazole 15 or 30 milligrams (mg), and participants who weigh >30 kg will be randomized to receive dexlansoprazole 30 or 60 mg.

All participants will be asked to take one capsule at the same time each day throughout the study. Parents/caregivers for participants ages 2 to 8 and participants ages 9 to 11 will be asked to record any time they have heartburn symptoms in an electronic diary.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is up to 16 weeks, which includes up to 4 weeks to screen for the study. Participants will make multiple visits to the clinic, plus a final phone call 5 to 10 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant (as age appropriate) and/or parent(s)/legal guardian is capable of understanding and complying with protocol requirements.
2. Prior to any study-specific procedures being performed, the appropriate informed consent and the assent form(s) (as applicable) must be signed and dated by parent(s) or legal guardian and by the participant respectively, if appropriate.
3. Has a medical history of symptoms of GERD for at least 3 months prior to Screening.
4. Has met the eDiary qualification criteria as assessed by the PGSDD, defined as hurting or burning in the stomach, chest, or throat on at least 3 of any 7 consecutive days during the Screening Period.
5. Has no evidence of erosive esophagitis (EE) according to the Los Angeles (LA) Classification of Esophagitis and, in the investigator's clinical judgment, the symptoms are suggestive of acid-related disease. A 24-hour pH-metry (with or without impedance) may be performed during Screening or within 6 months prior to Screening for similar symptoms as those identified during Screening if, in the investigator's judgment, this procedure would aid in the determination of whether the participant's symptoms are acid-related. An endoscopy performed within 1 week prior to signing screening informed consent and assent form (as applicable) is an acceptable replacement for the screening endoscopy if nonerosive GERD is confirmed, protocol-required biopsies were collected, and endoscopic pictures were obtained.
6. Is male or female and age 2 to 11 years, inclusive, at the time of screening informed consent.

Exclusion Criteria:

1. Has evidence of cardiovascular, pulmonary, central nervous system, hepatic, hematopoietic, renal, or metabolic disorder, severe allergy, asthma, or allergic skin rash that suggests any uncontrolled, clinically significant underlying disease or condition (other than the disease being studied), which may impact the ability of the participant to participate or potentially confound the study results.
2. Has a coexisting disease affecting the esophagus (eg, esophageal varices, scleroderma, viral or fungal infection, or esophageal stricture), history of radiation therapy or cryotherapy to the esophagus, caustic or physiochemical trauma such as sclerotherapy to the esophagus.
3. Has any findings in his/her medical history, physical examination, or safety clinical laboratory tests giving reasonable suspicion of underlying disease that might interfere with the conduct of the trial.
4. Has a history of hypersensitivity or allergies to dexlansoprazole or any component of the formulation of dexlansoprazole capsules, or any proton pump inhibitor (PPI) (including lansoprazole, omeprazole, rabeprazole, pantoprazole, or esomeprazole) or antacids.
5. Is required to take excluded medications or it is anticipated that the participant will require treatment with at least 1 of the disallowed concomitant medications during the study evaluation period.
6. Has a condition that may require inpatient surgery during the course of the study.
7. Has a known history of Barrett's esophagus with dysplastic changes in the esophagus.
8. Has a known history of eosinophilic esophagitis (EoE) or histologic findings suggestive of EoE (≥15 eosinophils per high-powered field [HPF]).
9. Has history of celiac disease, tests positive for tissue transglutaminase (tTG), antibody or confirmed disease by histology.
10. Has history of inflammatory bowel disease, or irritable bowel syndrome.
11. Has active gastric or duodenal ulcers within 4 weeks prior to Day -1. If present >4 weeks prior to Day -1, ulcers must not be present upon screening endoscopy.
12. Requires dilatation of esophageal strictures and/or strictures preventing passage of the endoscope during the screening endoscopy. Schatzki's ring (a ring of mucosal tissue near the lower esophageal sphincter) is acceptable.
13. A female participant who has reached menarche by Day -1.
14. Is known to be positive for the human immunodeficiency virus (HIV).
15. Has current or historical evidence of Zollinger-Ellison syndrome or other hypersecretory condition.
16. Has a history of gastric, duodenal, or esophageal surgery except simple oversew of an ulcer. A history of gastric tube and/or percutaneous endoscopic gastrostomy (PEG) placement is allowed.
17. Had an acute upper gastrointestinal hemorrhage within 4 weeks prior to endoscopy.
18. Has donated or lost >10% of the total blood volume, undergone plasmapheresis, or has had a transfusion of any blood product within 90 days prior to the first dose of study drug.
19. Has a known history of alcohol abuse or illegal drug use within the past 12 months prior to the first dose of study drug.
20. Has any screening abnormal laboratory value that suggests a clinically significant underlying disease or condition that may prevent the participant from entering the study; or the participant has: creatinine >1.5 mg/dL, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 times the upper limit of normal (×ULN), or total bilirubin >2.0 milligrams per deciliter (mg/dL) with AST/ALT elevated above the limits of normal values.
21. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study or may consent and assent (as applicable) under duress. Students of the institution/research facility who are under the supervision of, or in a subordinate role to, the investigator are also ineligible.
22. The participant, in the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.
23. Has participated in another clinical study (not including screening for Study TAK-390MR_205 [NCT02615184]) and/or has received any investigational compound within 30 days prior to Screening.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Days Without Hurting or Burning in the Stomach, Chest or Throat Over the 12 Weeks of Treatment | Up to 12 weeks
  Daily electronic diaries (eDiaries) will be completed which contain Pediatric Gastroesophageal Reflux Disease Symptom Daily Diaries (PGSDD) questionnaires that document presence or absence of hurting or burning in the stomach, chest or throat vomiting, regurgitation and trouble eating. Parents or caregivers of participants aged 2 to 8 years will complete the PGSDD (parent) in the eDiary for their child and participants aged 9 to 11 years will complete PGSDD (child) in the eDiary themselves. The eDiaries will be completed on a daily basis reflecting a continuous 24-hour period.

SECONDARY OUTCOMES:
Percentage of Days Without Hurting or Burning in the Stomach, Chest or Throat in Children Aged 9 to 11 Years Over the 12 Weeks of Treatment | Up to 12 weeks
  Daily eDiaries will be completed which contain PGSDD questionnaires that document presence or absence of hurting or burning in the stomach, chest or throat vomiting, regurgitation and trouble eating. Parents or caregivers of participants aged 2 to 8 years will complete the PGSDD (parent) in the eDiary for their child and participants aged 9 to 11 years will complete PGSDD (child) in the eDiary themselves. The eDiaries will be completed on a daily basis reflecting a continuous 24-hour period.
Percentage of Days Without Hurting or Burning in the Stomach, Chest or Throat in Children Aged 2 to 8 Years Over the 12 Weeks of Treatment | Up to 12 weeks
  Daily eDiaries will be completed which contain PGSDD questionnaires that document presence or absence of hurting or burning in the stomach, chest or throat vomiting, regurgitation and trouble eating. Parents or caregivers of participants aged 2 to 8 years will complete the PGSDD (parent) in the eDiary for their child and participants aged 9 to 11 years will complete PGSDD (child) in the eDiary themselves. The eDiaries will be completed on a daily basis reflecting a continuous 24-hour period.
Percentage of Days Without Vomiting Over the 12 Weeks of Treatment | Up to 12 weeks
  Daily eDiaries will be completed which contain PGSDD questionnaires that document presence or absence of hurting or burning in the stomach, chest or throat vomiting, regurgitation and trouble eating. Parents or caregivers of participants aged 2 to 8 years will complete the PGSDD (parent) in the eDiary for their child and participants aged 9 to 11 years will complete PGSDD (child) in the eDiary themselves. The eDiaries will be completed on a daily basis reflecting a continuous 24-hour period.
Percentage of Days Food Did Not Come Up from Stomach to Mouth Over the 12 Weeks of Treatment | Up to 12 weeks
  Daily eDiaries will be completed which contain PGSDD questionnaires that document presence or absence of hurting or burning in the stomach, chest or throat vomiting, regurgitation and trouble eating. Parents or caregivers of participants aged 2 to 8 years will complete the PGSDD (parent) in the eDiary for their child and participants aged 9 to 11 years will complete PGSDD (child) in the eDiary themselves. The eDiaries will be completed on a daily basis reflecting a continuous 24-hour period.
Percentage of Days Without Trouble Eating Over the 12 Weeks of Treatment | Up to 12 weeks
  Daily eDiaries will be completed which contain PGSDD questionnaires that document presence or absence of hurting or burning in the stomach, chest or throat vomiting, regurgitation and trouble eating. Parents or caregivers of participants aged 2 to 8 years will complete the PGSDD (parent) in the eDiary for their child and participants aged 9 to 11 years will complete PGSDD (child) in the eDiary themselves. The eDiaries will be completed on a daily basis reflecting a continuous 24-hour period.
Difference of the Median Percentage of Days Without Hurting or Burning in the Stomach, Chest, or Throat Over the 12 Weeks of Treatment Between the High Dose and the low Dose Within Each Weight Strata | Up to 12 weeks
  Daily eDiaries will be completed which contain PGSDD questionnaires that document presence or absence of hurting or burning in the stomach, chest or throat vomiting, regurgitation and trouble eating. Parents or caregivers of participants aged 2 to 8 years will complete the PGSDD (parent) in the eDiary for their child and participants aged 9 to 11 years will complete PGSDD (child) in the eDiary themselves. The eDiaries will be completed on a daily basis reflecting a continuous 24-hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (33):
- United States (17):
  - Childrens Center for Digestive Health Care, LLC, Mobile, Alabama
  - University of Utah/ Primary Childrens Hospital, San Francisco, California
  - Gastrointestinal Associates, PA, Centennial, Colorado
  - Envision Clinical Research, LLC, Miami, Florida
  - GI For Kids, Atlanta, Georgia
  - Strada Patient Care Center, Department of Pediatric Gastroenterology, Chicago, Illinois
  - Childrens Hospital of The Kings Daughters, Jackson, Mississippi
  - Maspons Pediatric Gastro, Manchester, New Hampshire
  - The University of Chicago, Cleveland, Ohio
  - Dartmouth-Hitchcock Manchester, Oklahoma City, Oklahoma
  - University of California San Francisco, Oklahoma City, Oklahoma
  - c/o Chelsea Campbell, RN, Knoxville, Tennessee
  - Vanderbilt University Medical Center,, Nashville, Tennessee
  - Oklahoma Pediatric Digestive Institute, El Paso, Texas
  - University Hospitals Cleveland Medical Center, Laredo, Texas
  - IMMUNOe Research Centers, Salt Lake City, Utah
  - National Research Centers, Norfolk, Virginia
- Canada (2):
  - Women and Children's Health Research Institute, Edmonton, Alberta
  - London Health Sciences Centre Children's Hospital, London, Ontario
- Colombia (3):
  - Hospital Universitario San Ignacio, Bogotá
  - Fundacion Valle del Lili, Cali
  - Centro Medico Imbanaco de Cali S.A, Cali
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Public Institution, Kaunas, LT
  - Vilnius University Hospital Santaros Klinikos, Public Institution, Vilnius, LT
- Mexico (5):
  - InspirePharma S. de R.L. de C.V., Monterrey, Nuevo León
  - Boca Clinical Trials Mexico S.C., Querétaro, Putumayo
  - Clinical Research Institute S.C., Tlalnepantla, State of Mexico
  - El Cielo Medical Center, Puebla City
  - SMIQ, S. DE R.L. DE C.V. Queretaro, Querétaro
- Poland (4):
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów, PL
  - In Vivo Osrodek Badan Klinicznych, Bydgoszcz
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Oddzial Gastroenterologii, Hepatologii, Zaburzen odzywiania i Pediatrii, Warsaw
  - Uniwersytecki Szpital Kliniczny im.Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b602f4db2bf003ab49d24?idFilter=%5B%22TAK-510-1001%22%2C%22TAK-935-18-002+%28OV935%29%22%2C%22TAK-935-1014%22%2C%22TAK-390MR_204%22%5D